CLINICAL TRIAL: NCT05234073
Title: Effects of a Four Weeks Social Emotional and Ethical Learning Training in Brazilian Public School Teachers: a Randomized Controlled Trial
Brief Title: Effects of a Four Weeks Social Emotional and Ethical Learning Training in Brazilian Public School Teachers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: Emory University (Other); GaiaMais (Unknown); Instituto Sidarta (Unknown); Universidade Federal do ABC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: HIAE_SEELT_BR
Record Dates: First submitted 2022-02-01; First posted 2022-02-10 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2022-10

CONDITIONS: Social Emotional Learning
Keywords: social emotional learning; teachers; well-being; stress
MeSH Terms: interventions — Waiting Lists

STUDY DESIGN:
Intervention Model Description: Teachers from the Public Education Network will be randomly assigned to paired classes. While one is attending the four-week online course classes and responding to the perceived mood states assessment questionnaires, the next class will be the control group and will be on hold until the next month answering the same emotional assessment questionnaires.
Who Masked: Participant
Masking Description: Teachers will be randomly distributed between the control and intervention groups without knowing which one they will participate in or the progress of the other class's processes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: A (first group to receive the intervention) (Experimental): The class will be instructed in the social emotional and ethical learning (SEELearning) for 4 weeks.
  Interventions: Behavioral: SEE Learning Online Training
- Experimental: B (second group to receive the intervention) (Experimental): This arm will not receive intervention in the first month and will receive SEE Learning after this period.
  Interventions: Behavioral: SEE Learning Online Training; Behavioral: Waiting list

INTERVENTIONS:
Behavioral: SEE Learning Online Training — This intervention includes classes about socioemotional learning theory and practice, topics related to ethics and well-being practices
Behavioral: Waiting list — This group will wait for one month to receive SEE Learning Online Training
  Arms: Experimental: B (second group to receive the intervention)

SUMMARY:
Social Emotional Learning (SEL) has gained importance in recent years and has been taught in several schools to support students in how to recognize and manage emotions, develop empathy, build cooperative relationships, solve problems effectively, and gain skills of communication. The objective of this study is to evaluate the effects of a training of 4-week Social Emotional and Ethical Learning on stress, well-being, socioemotional learning literacy, positive and negative affect, attention, and competent. This study will also assess the perception of teachers about training and its impact on their teaching skills and in personal life. Methods: Elementary and Secondary School Teachers public in Brazil (N = 1,500) will be invited to participate in the SEE training Learning. After signing the Free and Informed Consent Term, the they will be randomized into two groups A and B. Both groups will be before the experiment (T0), after one month (T1) and after two months (T2). ONE SEE Learning Training (SEELT) and B will be a checklist control group. Standby (WLC) for one month. After that, B will receive SEELT and A will not receive intervention, but will be guided to maintain the practices learned. RESULTS EXPECTED: The groups after receiving the SEELT should present better results relating to their socio-emotional skills, stress management, increase in well-being and knowledge about these skills, are still so, better prepared to teach their students.

ELIGIBILITY:
Inclusion Criteria:

* Teachers from the public schools in Brazil

Exclusion Criteria:

-

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1500 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Change in stress | 1 month
  The authors will evaluate stress using the 10-item perceived stress scale. Higher values means worse stress.
  2. change in attention The authors will apply the Perceived Stress Scale
Change in well-being perception | 1 month
  The authors will evaluate well-being using the World Health Organization 5-item well-being index. Higher scores means better well-being.
Understanding of the application of socio-emotional and ethical learning | 1 month
  Questionnaire on Knowledge about Socioemotional Learning and Ethics. This is a 0 to 10 score questionnaire. Higher scores means better understanding in the topic.

SECONDARY OUTCOMES:
Effectiveness of content learning and training appreciation | 1 month
  Qualitative interviews in focus groups will be carried out among the participants
change in positive and negative affect (PANAS) | 1 month
  The authors will apply Positive and Negative Affect Scale (PANAS). Higher scores in negative affect means worse affective state and higher scores in positive affect means better affective state.
Perception of Stress, Well-Being, Attention, Frustration, Motivation in the last week | 1 month
  the author will aply "Questionary of Perception of Stress, Well-Being, Attention, Frustration, Motivation in the Last Week". Each item will be answered in a 0 to 10 item scale. The minimum value is 0 and the maximum is 10. Higher scores in stress and frustration are worse scores. Higher scores in well-being, attention and motivation are better scores in the questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Israelita Albert Einstein, São Paulo, Brazil